CLINICAL TRIAL: NCT06145373
Title: An Open-label, Single-arm Treatment Study to Investigate the Safety and Tolerability of Switching From Emicizumab to Fitusiran Prophylaxis in Male Participants Aged ≥12 Years of Age With Severe Hemophilia A, With or Without Inhibitors
Brief Title: A Study to Test a Medicine (Fitusiran) for Preventing Bleeds in People With Severe Hemophilia Who Previously Received Preventive Treatment With Emicizumab
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFY17741; 2022-502414-84 (Registry Identifier: CTIS); U1111-1280-7227 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — fitusiran; emicizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- fitusiran (Experimental): The pre-fitusiran treatment period is defined as the transition period up to the first fitusiran administration. Participants will receive on demand or prophylactic treatment with intravenous clotting factor concentrates (IV CFCs) or bypassing agents (BPAs) from Month-2 until Day 1.
  Fitusiran treatment period: Participants will receive subcutaneous (SC) fitusiran prophylaxis once every 2 months (Q2M) or once monthly (QM) from Day 1 until Month18.
  Participants may receive IV antithrombin concentrate (ATIIIC) upon investigator's judgement.
  AT FU period: Participants will be followed up until AT activity levels recover to at least 60% (per central laboratory).
  In case of bleeding events participants will receive IV CFCs or BPAs. Participants may receive IV ATIIIC upon investigator's judgement.
  Interventions: Drug: Fitusiran (SAR439774); Biological: Clotting factor concentrates (CFC) or bypassing agents (BPA); Biological: Antithrombin concentrate (ATIIIC); Biological: Emicizumab

INTERVENTIONS:
Drug: Fitusiran (SAR439774) — Pharmaceutical form:Solution for injection-Route of administration:Subcutaneous (SC) injection
  Other Names: SAR439774, Qfitlia®
Biological: Clotting factor concentrates (CFC) or bypassing agents (BPA) — Pharmaceutical form: Solution for injection-Route of administration: Intravenous (IV) injection
Biological: Antithrombin concentrate (ATIIIC) — Pharmaceutical form:Solution for injection-Route of administration:Intravenous (IV) injection
Biological: Emicizumab — Pharmaceutical form:Solution for injection-Route of administration:SC injection

SUMMARY:
This is an exploratory, single group, Phase 4, study to assess treatment with fitusiran prophylaxis after switching from emicizumab prophylaxis.

This study aims to evaluate the safety and tolerability of switching to fitusiran after a transition period from the last dose of emicizumab. The study will be conducted in male participants with severe hemophilia A, with or without inhibitors, aged ≥12 years, who were previously receiving emicizumab prophylaxis.

Study details include:

* The study duration will be up to approximately 28 months:

  * There will be an approximately 2-month screening period.
  * There will be an approximately 2-month period before fitusiran treatment starts (pre-fitusiran treatment period)
  * The fitusiran treatment duration will be up to 18-months (fitusiran treatment period)
  * The antithrombin (AT) follow-up (FU) period will be approximately 6 months after the last dose of fitusiran (during which the AT activity level will be monitored at approximately monthly intervals following the final fitusiran dose until AT activity levels return to at least 60%).
* The study site visits are scheduled at monthly/ every 2 months intervals of 28 days (4 weeks) / 56 days (8 weeks), respectively, during the fitusiran treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male participants must be ≥12 years of age inclusive, at the time of signing the informed consent
* Diagnosis of severe congenital hemophilia A (FVIII < 1%) as evidenced by a central laboratory measurement at screening or documented medical record evidence.

  * Inhibitor titer of ≥0.6 BU/mL at Screening, or
  * Inhibitor titer of <0.6 BU/mL at Screening with medical record evidence of 2 consecutive titers ≥0.6 BU/mL, or
  * Inhibitor titer of <0.6 BU/mL at Screening with medical record evidence of anamnestic response.
* Participants who are currently on the full labeled dose of emicizumab prophylaxis, irrespective of inhibitor/non-inhibitor status.
* Signed informed consent/assent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known coexisting bleeding disorders
* History of antiphospholipid antibody syndrome.
* History of arterial or venous thromboembolism, atrial fibrillation, significant valvular disease, myocardial infarction, angina, transient ischemic attack, or stroke. Participants who have experienced thrombosis associated with indwelling venous access may be enrolled.
* Presence of clinically significant liver disease
* Current or prior participation in a fitusiran trial
* Current or prior participation in a gene therapy trial
* AT activity <60% at Screening, as determined by central laboratory measurement
* Coexisting thrombophilic disorder - Hepatitis C virus antibody positive, except participants who have negative Hepatitis C viral load and no evidence of cirrhosis
* Presence of acute hepatitis, ie, hepatitis A, hepatitis E.
* Presence of acute or chronic hepatitis B infection
* Known to be HIV positive with CD4 count <200 cells/μL.
* Reduced renal function

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-09-19 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse events (AEs) during the fitusiran treatment | From Day 1 up to Month 4
  Incidence, severity, and seriousness, of AEs occurred during fitusiran treatment period will be reported

SECONDARY OUTCOMES:
The peak thrombin generation (TG) - pre fitusiran treatment | From Month -2 up to Day 1
  Central laboratory assessments (peak TG) will be reported for pre-fitusiran period
The peak TG during fitusiran treatment | From Day 1 up to Month 4
  Central laboratory assessments (peak TG) will be reported for fitusiran treatment period
The antithrombin (AT) levels during pre-fitusiran treatment | From Month -2 up to Day 1
  Central laboratory assessments (AT) will be reported for pre-fitusiran treatment period
The AT levels during fitusiran prophylaxis | From Day 1 up to Month 4
  Central laboratory assessments (AT) will be reported for fitusiran treatment
Emicizumab concentrations in plasma | Up to Month 4 of fitusiran treatment
  Emicizumab concentrations in plasma will be reported
Number of participants with AEs from Day 1 to Month 18 of fitusiran treatment | From Day 1 up to Month 18
  Incidence, severity, and seriousness of AEs will be reported
Change in participants' overall treatment satisfaction during the fitusiran treatment period assessed via the Treatment Satisfaction Questionnaire for Medication (TSQM-9) domain scores | From approximately Month -2 to Month 19 [end of study (EoS) visit]
  The three domains of effectiveness, convenience, and global satisfaction will be reported
Participants' treatment preferences (via the Preference Questionnaire) | At Month 12
  The Preference questionnaire Data will be reported
Change in adult participants' pain intensity during the fitusiran treatment period over time | From approximately Month - 2 to Month 19 (EoS) visit
  The PROMIS (Patient-Reported Outcomes Measurement Information System) Pain Intensity 3a v2.0 consists of three items measuring the worst, average, and current intensity of pain with a recall period of 7 days. Each question has five response options ranging from one ('no pain') to five ('very severe').
  Adult participants (age ≥ 18 years) will self-complete the PROMIS Pain Intensity 3a v2.0 questionnaire.
Change in adolescent participants' pain intensity during the fitusiran treatment period over time | From approximately Month - 2 to Month 19 (EoS) visit
  The PROMIS Pediatric Numeric Rating Scale v.1.0 - Pain Intensity 1a consists of one item measuring the average intensity of pain with a recall period of 7 days. The question has ten response options ranging from one ('no pain') to ten ('worst pain').
  Adolescent participants (age ≥12 years and <17 years) will self-complete the PROMIS Pediatric Pain Intensity 1a v.1.0.
Change in participants' physical functioning and physical activity during the fitusiran treatment period (via the International Physical Activity Questionnaire [IPAQ]) over time | From approximately Month - 2 to Month 19 (EoS) visit
  Participants' physical functioning and physical activity data during the fitusiran treatment period will be collected via the International Physical Activity Questionnaire and reported
Change in participants' joint health (via the Hemophilia Joint Health Score [HJHS]) during the fitusiran treatment period over time | From approximately Month - 2 to Month 19 (EoS) visit
  HJHS during the fitusiran treatment period will be reported
Annualized Bleeding Rate (ABR) while receiving fitusiran prophylaxis | From Month 4 up to Month 18 (14-month extension period)
  The frequency of treated bleeding episodes will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Children's Hospital Los Angeles- Site Number : 8400005, Los Angeles, California, United States
- Investigational Site Number : 1580001, Taipei, Podlaskie, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: SFY17741 Plain Language Results Summaries — https://www.trialsummaries.com/Study/StudyDetails?id=25530&tenant=MT_SNY_9011